CLINICAL TRIAL: NCT04138758
Title: Effectiveness and Safety of Maintenance Treatment With Combination of Tiotropium and Olodaterol in Comparison to Maintenance Treatment With a Combination of Inhaled Corticosteroids and Long-acting β2 Agonists in COPD Patients
Brief Title: Comparative Effectiveness and Safety of Tiotropium and Olodaterol in Comparison to LABA/ICS
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0093
Record Dates: First submitted 2019-10-23; First posted 2019-10-24 (Actual); Results first posted 2020-11-30 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients initiating Tiotropium+Olodaterol therapy
  Interventions: Drug: Tiotropium bromide + Olodaterol
- Patients initiating Long-acting beta agonist/inhaled corticosteroid therapy
  Interventions: Drug: LABA/ICS

INTERVENTIONS:
Drug: Tiotropium bromide + Olodaterol — Tiotropium bromide + Olodaterol
  Groups: Patients initiating Tiotropium+Olodaterol therapy
Drug: LABA/ICS — Long-acting beta2-agonist and Inhaled corticosteroids (LABA and ICS)
  Groups: Patients initiating Long-acting beta agonist/inhaled corticosteroid therapy

SUMMARY:
The primary objective is to compare the effectiveness of maintenance therapy initiation with the combination treatment Tiotropium and Olodaterol (Olo+Tio) compared with LABA/ICS combination in COPD as the time to the first COPD exacerbation.

Secondary objectives are to compare patients treated with Tio+Olo and patients treated with LABA/ ICS combination.

ELIGIBILITY:
Inclusion Criteria:

1. At least one prescription for Tio+Olo combined inhaler or a LABA/ICS combined inhaler between 1 January 2013 and 31 March 2019.

   1. The first dispensing of either Tio+Olo or LABA/ICS combined inhaler will be defined as the index date.
   2. For the main analyses, only fixed dose combination (FDC) inhalers will be included. Sensitivity analyses will also accept free combinations of LABA/ICS.
2. At least one diagnosis of COPD at any time prior to the index date.
3. At least one year of continuous medical and pharmacy health plan eligibility prior to the index date will be required to allow a baseline period for the covariates and identification of new use of the study drugs.

Exclusion Criteria:

1. To increase the likelihood of a true diagnosis of COPD, we will exclude:

   1. All patients less than 40 years of age on the index date, and
   2. All patients with a diagnosis of asthma in the year prior to the index date
2. To limit the population to those without severe lung compromise outside of COPD, we will exclude individuals with lung cancer, interstitial lung disease, or lung transplant identified at any time prior to the index date
3. To restrict the cohort to new users of Tio+Olo or LABA/ICS, we will exclude any individual with use of either Tio+Olo, LABA/ICS, or LABA/LAMA/ICS combination therapy in free or fixed form for at least one year prior to the index date.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with COPD inititated with Tio+Olo in comparison to patients treated with ICS/LABA/LAMA
Sampling Method: Non-Probability Sample
Enrollment: 42953 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- HealthCore, Inc., Watertown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Quint JK, Montonen J, Esposito DB, He X, Koerner L, Wallace L, de la Hoz A, Miravitlles M. Effectiveness and Safety of COPD Maintenance Therapy with Tiotropium/Olodaterol versus LABA/ICS in a US Claims Database. Adv Ther. 2021 May;38(5):2249-2270. doi: 10.1007/s12325-021-01646-5. Epub 2021 Mar 15. PMID 33721209
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this cohort study, administrative data from the HealthCore Integrated Research Database (US, HIRD, Jan 2013 - March 2019) were used to identify and compare new users of Tio+Olo (Tiotropium and Olodaterol) with new users of LABA/ICS (Long-acting Beta2-Agonists/Inhaled Corticosteroids) combination therapy with respect to safety and effectiveness.
Pre-assignment Details: Only subjects that met all inclusion and none of the exclusion criteria were included. two cohorts (Initiators of Tiotropium + Olodaterol and patients receiving Long-acting beta agonist / inhaled corticosteroid) were established. The cohorts after propensity score matching were used for the analyses
Groups:
- Tiotropium + Olodaterol: Cohort of patients with Chronic Obstructive Pulmonary Disease (COPD) derived from administrative data from the HealthCore Integrated Research Database (HIRD, January 2013 - March 2019), who initiated fixed dose combination (FDC) inhaler treatment of Tiotropium and Olodaterol, with the first prescription defined as the index date. Following the index date participants were followed for up to one year.
- Long-acting Beta Agonist / Inhaled Corticosteroid Therapy: Cohort of patients with Chronic Obstructive Pulmonary Disease (COPD) derived from administrative data from the HealthCore Integrated Research Database (HIRD, January 2013 - March 2019), who initiated long-acting beta agonist / inhaled corticosteroid therapy, with the first prescription defined as the index date. Following the index date participants were followed for up to one year.
Period: Overall Study
Arm/Group | Tiotropium + Olodaterol | Long-acting Beta Agonist / Inhaled Corticosteroid Therapy
Started | 2600 | 40353
Completed | 2600 | 40353
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Propensity score weighted populations of patients with Chronic Obstructive Pulmonary Disease (COPD) derived from the HealthCore Integrated Research Database (HIRD, January 2013 - March 2019), who initiated fixed dose combination (FDC) inhaler treatment of Tiotropium and Olodaterol or long-acting beta agonist / inhaled corticosteroid therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium + Olodaterol | Long-acting Beta Agonist / Inhaled Corticosteroid Therapy | Total
Number analyzed (Participants) | 2600 | 40353 | 42953
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10.3) | 64.8 (11.5) | 64.81 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1415 | 21994 | 23409
  Male | 1185 | 18359 | 19544
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Description: Incidence rate of Chronic Obstructive Pulmonary Disease (COPD) exacerbation after cohort entry. The event was defined as follows:
  Severe exacerbation: Hospitalization with a principal discharge diagnosis of COPD.
  or Moderate exacerbation: An emergency department (ED) visit with a discharge diagnosis of COPD, or, an antibiotic for a respiratory condition dispensed the same day as an oral corticosteroid.
Time Frame: From cohort entry (index date) until the occurrence of a hospitalization for COPD (severe exacerbation), ED visit for COPD or prescription of an antibiotic and oral corticosteroid on the same day (moderate exacerbation). Up to one year after cohort entry.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Events per 1,000 Person-days
Arm/Group | Tiotropium + Olodaterol | Long-acting Beta Agonist / Inhaled Corticosteroid Therapy
Number analyzed (Participants) | 2600 | 40353
Events per 1,000 Person-days | 1.63 [1.47 to 1.81] | 2.43 [2.37 to 2.49]
Statistical Analysis 1: Comparison: Tiotropium + Olodaterol vs Long-acting Beta Agonist / Inhaled Corticosteroid Therapy; Cox proportional hazard regression models were used to assess the effect of Tiotropium + Olodaterol combination versus the Long-acting beta agonist / inhaled corticosteroid therapy combination on the risk of a first COPD exacerbation; Test type: Other; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.68 to 0.85] — Hazard Ratio lower than 1 favors Tiotropium + Olodaterol

2. Secondary Outcome: Incidence Rate of First Hospitalization for Community-acquired Pneumonia
Description: Incidence rate of first hospitalization for community-acquired pneumonia (serious pneumonia). Pneumonia was defined using ICD-9-CM diagnoses and ICD-10 diagnosis codes.
Time Frame: From cohort entry (index date) until the occurrence of first hospitalization for community-acquired pneumonia (serious pneumonia). Up to one year after cohort entry.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: events per 1,000 Person-days
Arm/Group | Tiotropium + Olodaterol | Long-acting Beta Agonist / Inhaled Corticosteroid Therapy
Number analyzed (Participants) | 2600 | 40353
events per 1,000 Person-days | 0.23 [0.18 to 0.30] | 0.34 [0.32 to 0.37]
Statistical Analysis 1: Comparison: Tiotropium + Olodaterol vs Long-acting Beta Agonist / Inhaled Corticosteroid Therapy; Cox proportional hazard regression models were used to assess the effect of Tiotropium + Olodaterol combination versus the Long-acting beta agonist / inhaled corticosteroid therapy combination on the risk of first hospitalization for community-acquired pneumonia; Test type: Other; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.57 to 0.97] — Hazard Ratio lower than 1 favors Tiotropium + Olodaterol

3. Secondary Outcome: Incidence Rate of the First Date of a Pharmacy Dispensing Indicating Escalation (Original Case Definition) to Triple Therapy
Description: Incidence rate of the first date of a pharmacy dispensing indicating escalation to triple therapy, (i.e., addition of Inhaled Corticosteroids to Tiotropium and Olodaterol or a Long-acting Muscarinic Antagonists to long-acting beta agonist / inhaled corticosteroid therapy).
Time Frame: From cohort entry (index date) until the escalation, up to one year after cohort entry.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: events per 1,000 Person-days
Arm/Group | Tiotropium + Olodaterol | Long-acting Beta Agonist / Inhaled Corticosteroid Therapy
Number analyzed (Participants) | 2600 | 40353
events per 1,000 Person-days | 0.54 [0.46 to 0.64] | 2.90 [2.84 to 2.97]
Statistical Analysis 1: Comparison: Tiotropium + Olodaterol vs Long-acting Beta Agonist / Inhaled Corticosteroid Therapy; Test type: Other — Cox proportional hazard regression models were used to assess the effect of Tiotropium + Olodaterol combination versus the Long-acting beta agonist / inhaled corticosteroid therapy combination on the risk of escalation; Hazard Ratio (HR) = 0.23, 95% CI 2-sided [0.19 to 0.27] — Hazard Ratio lower than 1 favors Tiotropium + Olodaterol

4. Secondary Outcome: Incidence Rate of the First Date of a Pharmacy Dispensing Indicating Escalation (Alternative Case Definition) to Triple Therapy
Description: Incidence rate of the first date of a pharmacy dispensing indicating escalation to triple therapy.
  Based on feedback from clinical experts during review of study results, an alternative post-hoc definition was also assessed in which initiation of any treatment including simultaneous LABA (long-acting beta agonist) /LAMA (Long-acting Muscarinic Antagonists) /ICS (inhaled corticosteroid therapy) use in free or fixed combination was counted as an outcome.
Time Frame: From cohort entry (index date) until the escalation, up to one year after cohort entry.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: events per 1,000 Person-days
Arm/Group | Tiotropium + Olodaterol | Long-acting Beta Agonist / Inhaled Corticosteroid Therapy
Number analyzed (Participants) | 2600 | 40353
events per 1,000 Person-days | 0.57 [0.48 to 0.67] | 3.14 [3.08 to 3.21]
Statistical Analysis 1: Comparison: Tiotropium + Olodaterol vs Long-acting Beta Agonist / Inhaled Corticosteroid Therapy; Cox proportional hazard regression models were used to assess the effect of Tiotropium + Olodaterol combination versus the Long-acting beta agonist / inhaled corticosteroid therapy combination on the risk of escalation; Test type: Other; Hazard Ratio (HR) = 0.22, 95% CI 2-sided [0.19 to 0.26] — Hazard Ratio lower than 1 favors Tiotropium + Olodaterol

5. Secondary Outcome: Incidence Rate of Any Element of a Composite Outcome Including Exacerbation, Hospitalization for Pneumonia, or Escalation (Original Case Definition) to Triple Therapy
Description: Incidence rate of any element of a composite outcome including exacerbation, hospitalization for pneumonia, or escalation (original case definition) to triple therapy.
  Exacerbation was defined as follows: Severe exacerbation: Hospitalization with a principal discharge diagnosis of COPD. Moderate exacerbation: An emergency department (ED) visit with a discharge diagnosis of COPD, or, an antibiotic for a respiratory condition dispensed the same day as an oral corticosteroid.
  Pneumonia was defined using ICD-9-CM diagnoses and ICD-10 diagnosis codes. Escalation was defined as the addition of Inhaled Corticosteroids to Tiotropium and Olodaterol or a Long-acting Muscarinic Antagonists to long-acting beta agonist / inhaled corticosteroid therapy.
Time Frame: From cohort entry (index date) until exacerbation, hospitalization (for community-acquired pneumonia) or escalation, up to one year after cohort entry.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: events per 1,000 Person-days
Arm/Group | Tiotropium + Olodaterol | Long-acting Beta Agonist / Inhaled Corticosteroid Therapy
Number analyzed (Participants) | 2600 | 40353
events per 1,000 Person-days | 2.14 [1.96 to 2.34] | 5.45 [5.36 to 5.54]
Statistical Analysis 1: Comparison: Tiotropium + Olodaterol vs Long-acting Beta Agonist / Inhaled Corticosteroid Therapy; Cox proportional hazard regression models were used to assess the effect of Tiotropium + Olodaterol combination versus the Long-acting beta agonist / inhaled corticosteroid therapy combination on the risk of any element of a composite outcome including exacerbation, hospitalization for pneumonia, or escalation; Test type: Other; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.42 to 0.51] — Hazard Ratio lower than 1 favors Tiotropium + Olodaterol

6. Secondary Outcome: Incidence Rate of Any Element of a Composite Outcome Including Exacerbation, Hospitalization for Pneumonia, or Escalation (Alternative Case Definition) to Triple Therapy
Description: Incidence rate of any element of a composite outcome including exacerbation, hospitalization for pneumonia, or escalation (alternative case definition) to triple therapy.
  Exacerbation was defined as follows: Severe exacerbation: Hospitalization with a principal discharge diagnosis of COPD. Moderate exacerbation: An emergency department (ED) visit with a discharge diagnosis of COPD, or, an antibiotic for a respiratory condition dispensed the same day as an oral corticosteroid.
  Pneumonia was defined using ICD-9-CM diagnoses and ICD-10 diagnosis codes. Escalation was defined as the initiation of any treatment including simultaneous LABA (long-acting beta agonist) /LAMA (Long-acting Muscarinic Antagonists) /ICS (inhaled corticosteroid therapy) use in free or fixed combination.
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: events per 1,000 Person-days
Arm/Group | Tiotropium + Olodaterol | Long-acting Beta Agonist / Inhaled Corticosteroid Therapy
Number analyzed (Participants) | 2600 | 40353
events per 1,000 Person-days | 2.16 [1.98 to 2.37] | 5.67 [5.58 to 5.77]
Statistical Analysis 1: Comparison: Tiotropium + Olodaterol vs Long-acting Beta Agonist / Inhaled Corticosteroid Therapy; [analysis description as in outcome 5, analysis 1]; Test type: Other; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.41 to 0.49] — Hazard Ratio lower than 1 favors Tiotropium + Olodaterol

ADVERSE EVENTS:
Description: As this is a non-interventional study with secondary use of data retrieved from a US health claims database, safety monitoring and safety reporting on an individual case level is not applicable.
  Total number of participants at risk is 0 since adverse events were not planned to be collected and reported for this study.
Arm/Group | Tiotropium + Olodaterol | Long-acting Beta Agonist / Inhaled Corticosteroid Therapy
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT04138758/Prot_SAP_000.pdf